CLINICAL TRIAL: NCT05732506
Title: Safety Evaluation of Edoxaban in Elderly Patients With Frailty Criteria
Status: Completed | Type: Observational
Sponsor: Galaxia Empírica (Network)
Responsible Party: Sponsor
Other Study IDs: EDO-FRAG-001
Record Dates: First submitted 2023-02-07; First posted 2023-02-17 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Auricular Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Elderly patients diagnosed with nonvalvular atrial fibrillation who meet the frailty criteria and who had been receiving anticoagulant treatment with Edoxaban for no more than 6 months prior to inclusion in the study.
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — There are not intervention.
  Other Names: Lixiana

SUMMARY:
The aim of the present study is to prospectively evaluate the safety of Edoxaban.

DETAILED DESCRIPTION:
The aim of the present study is to prospectively evaluate the safety of Edoxaban in daily clinical practice in Spain in elderly patients with nonvalvular atrial fibrillation who meet the criteria for frailty and who have been prescribed the drug recently (<6 months prior to inclusion).

The study will provide us with a clear and real-life picture of bleeding and ischemic complications and possible treatment interruptions with Edoxaban in real life and in a large subgroup, although underrepresented in the studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients 75 years of age or older with a diagnosis of NVAF.
* Patients in whom treatment had been started in the 6 months prior to enrollment in the study with Edoxaban for prevention of stroke and systemic embolism after diagnosis of NVAF and according to the drug's technical data sheet.
* Frailty criteria according to the FRAIL scale (score of 3 to 5 points).
* Written informed consent to participate in the study prior to any intervention.

Exclusion Criteria:

* Creatinine clearance according to the CKD-EPI formula less than 15 ml/min/m2
* Moderate or severe hepatic insufficiency (Defined as grade B or C of the Child-Pugh classification.
* Contraindication to receive Edoxaban according to the Technical Data Sheet.
* Participation in any clinical drug trial in the 2 months prior to the initial visit.
* Absence of recorded patient or treatment information.
* Surgical or percutaneous occlusion of the left atrial appendage or intention to perform such intervention at the time of inclusion.
* Any circumstance that, in the opinion of the investigator, affects patient follow-up (including life expectancy of less than two years or inability to perform follow-up).
* Persons who are legally incapacitated or unable to understand informed consent.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will consist of patients ≥75 years diagnosed with NVAF who meet frailty criteria and who have been receiving anticoagulation therapy with Edoxaban for no more than 6 months prior to study inclusion according to AEMPS recommendations and the summary of product characteristics.
Sampling Method: Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Major bleeding. | 12 months
  Proportion of patients who had a major bleeding during the 12 months of follow-up.

SECONDARY OUTCOMES:
Stroke or systemic embolism. | 12 months
  Proportion of patients who suffered stroke or systemic embolism during the 12 months of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro Hermida Ameijeiras, Principal Investigator
Locations (35):
- Spain (35):
  - Complejo Hospitalario Universitario de A Coruña, A Coruña, A Coruña
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, A Coruña
  - Hospital Universitario de Áraba, Vitoria-Gasteiz, ALAVA
  - Hospital Universitario Nuestra Señora del Perpetuo Socorro, Albacete, Albacete
  - Hospital Vega Baja, Alicante, Alicante
  - Hospital Universitario del Vinalopó, Elche, Alicante
  - Hospital Perpetuo Socorro, Badajoz, Badajoz
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de Sant Juan Despí, Sant Joan Despí, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de La Plana, Ciudad Real, Castellón
  - Hospital San Pedro de Alcántara, Cáceres, Cáceres
  - Hospital Virgen del Puerto Plasencia, Plasencia, Cáceres
  - Hospital Universitario Puerto Real, Puerto Real, Cádiz
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, Galicia
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Universitario Doctor José Molina Orosa, Arrecife, Las Palmas
  - Hospital Universitario de León, León, León
  - Hospital del Bierzo, Ponferrada, León
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital Universitario Puerta De Hierro, Majadahonda, Madrid
  - Hospital Infanta Sofia, San Sebastián de los Reyes, Madrid
  - Hospital Regional Universitario de Málaga, Málaga, Málaga
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Monte Naranco, Oviedo, Principality of Asturias
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Santa Cruz De Tenerife
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided